CLINICAL TRIAL: NCT01380171
Title: Primary Palatoplasty in Pediatric Patients - A Retrospective Review of Surgical Outcomes
Status: Completed | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: John Riski, PhD, Children's Healthcare of Atlanta
Other Study IDs: 06-196
Record Dates: First submitted 2010-05-24; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Cleft Lip; Cleft Palate
MeSH Terms: conditions — Cleft Lip; Cleft Palate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cleft lip/palate: Patients who have had surgical intervention for cleft lip/palate since 1998 at Children's Healthcare of Atlanta at the Center for Craniofacial Disorders

SUMMARY:
Children who are born with cleft palate need surgery in order to correct the problem. The surgery is needed because the defect allows food to leak into the nose. It also causes the patient to be unable to speak correctly, producing a problematic nasal sound. Sometimes the first surgery does not completely correct the problem and a second surgery is needed. Looking at the records of patients who have had corrective surgeries done in the past would allow the surgeons to improve their success rate and reduce the need for secondary surgeries. It would also create greater patient safety and reduce cost for families.

DETAILED DESCRIPTION:
Background and Purpose:

Children born with cleft palate require surgical correction in order to prevent nasal regurgitation of food and in order to create normal palate function for speech. Uncorrected, speech is hypernasal and unintelligible. Normal speech has very few sounds that are normally nasal. In English, there are only three, "m" as in "Mama", "n" as in "no", and "ng" as in "ring". The remaining 43 sounds in English are made with the soft palate (or velum) closing off the nasopharynx, and projecting speech orally. The goal for surgical separation of the nose and mouth at the hard palate (palatoplasty) is to create a complete separation of the nose and mouth at the hard palate and a functioning soft palate that can open and close the nasopharynx appropriately for speech sound.

Unfortunately, primary closure of the palate is not completely successful in all patients. In some patients, an opening (fistula) remains in the (anterior) hard palate allowing food and speech to leak through the nose. A second problem is that the (posterior) soft palate may not be long enough or move far enough to close off the nasopharynx. This is called a velopharyngeal incompetence. These patients may also suffer from nasal regurgitation and hypernasal, unintelligible speech. Both palatal fistula and velopharyngeal incompetence will require secondary surgery. Any information gained from review of surgical outcomes of the primary palatoplasty might improve surgical success and reduce the number of secondary surgeries required. This would reduce possible morbidity to the patient and expense to the families.

The purpose of this review will be to evaluate the outcome of the palatoplasty children and follow through the Center for Craniofacial Disorders at Children's Healthcare of Atlanta on the Scottish Rite campus. The investigators will evaluate for the occurence of palatal fistula and velopharyngeal incompetence.

Summary of Procedures:

General Procedures: The clinical databases at the Center for Craniofacial Disorders will be evaluated Locations Involved: The Center for Craniofacial Disorders is at Children's Healthcare of Atlanta and is on the Scottish Rite campus Number of Subjects: 1295 patients have been treated since 1998.

Potential Risks:

There are no physical, psychological, or financial risks to the patients.

Due to the nature of this records review study, information collected in this study will contain Protected Health Information (PHI) on subjects. There is the potential risk of unintentional disclosure of this information. However, certain steps will be followed in this study to minimalize PHI disclosure to help protect the subjects' privacy and confidentiality. Patient confidentiality wil be protected since the databases are on secure servers within the Children's network. The databases are password-protected and are accessible only to clinicians entering clinical notes and approved researchers. Other than institutions required by law to have access to research records, only authorized research staff will have access to the research database associated with the study. Furthermore, no data will be identifiable to study subjects, as each subject will be assigned a unique study number when entered into a database. If published or presented, no identifying features will be provided.

Potential Benefits:

There might be no immediate benefit to the patients whose records are evaluated. There is potential benefit to future patients seen at the Center. Evaluation of surgical outcomes might identify potential hazards that reduce the effectiveness of surgery. Efforts can be made to avoid these hazards in the future. The investigators might also find that certain surgical techniques or ages at surgery lead to better outcomes. Surgical protocol could be modified with the potential of improvement of surgical outcomes in the future.

Informed Consent Process:

Due to the nature of this retrospective records review study, informed consent from the subjects is not required and a Request for Waiver of Authorization was submitted. This research involves no more than minimal risk to the subjects, as there will be no subject contact and only the subjects' data will be utilized in the conduct of the research. There is the minimal risk of a breach in confidentiality with the subjects' PHI being disclosed, however, a procedure is in place for the protection of any collected PHI. The waiver of informed consent will not adversely affect the rights and welfare of the subject as this research does not change their standard of care and their confidentiality rights will be respected. This research could not be practicably carried out without the waiver of the informed consent as it is a retrospective chart review study where subject data is needed to meet the objectives of the study and consent cannot be practicably obtained from the patients. Whenever appropriate, the subjects will be provided with additional pertinent information after participation, however, in this case, the subjects' standard of care will not be affected so there will be no need for contact with subjects. The Request for Waiver of Authorization outlines the types of PHI that will be collected, protection and destruction plan for PHI, assurances against PHI re-disclosure, and the need for collection of PHI in order to conduct the study.

ELIGIBILITY:
Inclusion Criteria:

* Children operated on by surgeons at the Center for Craniofacial Disorders
* Have a diagnosis of cleft lip/palate
* Children with a syndrome in addition to cleft lip/palate will be evaluated in a different category

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1295 patients with cleft lip/palate that have been treated since 1998 at the Center for Craniofacial Disorders at Children's Healthcare of Atlanta on the Scottish Rite campus.
Sampling Method: Non-Probability Sample
Enrollment: 1295 (Actual)
Dates: Start 2007-02; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Riski, PhD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta at Scottish Rite, Atlanta, Georgia, United States

REFERENCES:
- See also: Children's Healthcare of Atlanta's main public website — http://www.choa.org